CLINICAL TRIAL: NCT04462393
Title: Characteristics and Outcomes of Patients Admitted to Swedish Intensive Care Units for COVID-19 During the First 60 Days of the 2020 Pandemic
Brief Title: Characteristics and Outcomes of Patients Admitted to Swedish Intensive Care Units for COVID-19
Status: Active, not recruiting | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: Region Östergötland (Other)
Responsible Party: Principal Investigator, Michelle Chew, Professor, Linkoeping University
Other Study IDs: SweCOVID
Record Dates: First submitted 2020-07-06; First posted 2020-07-08 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; Critical Illness
MeSH Terms: conditions — COVID-19; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Admission to ICU for COVID-19 — All patients admitted to Swedish ICUs with COVID-19 between 6 Mar - 6 May 2020

SUMMARY:
This is a registry-based cohort study of all adult patients (≥18 years) admitted to Swedish Intensive Care Units with confirmed SARS-CoV-2 infection and COVID-19 disease during the first 2 months of the 2020 pandemic.

The main goal is to describe demographic characteristics, coexisting conditions, treatments and outcomes among critically ill patients with COVID-19. A secondary goal is to identify independent risk factors associated with increased mortality for these patients.

Data regarding baseline characteristics including comorbidities, intensive care treatments and outcomes will be extracted. ICU lengths of stay and 30-day mortalities will be calculated. The primary outcome is 30-day all-cause mortality. THIS PART OF THE STUDY HAS BEEN COMPLETED.

UPDATE 26 Feb 2022:

Characteristics and outcomes of 'first wave' patients admitted to Swedish ICUs was published in Eur J Anaesthesiol. 2021 Apr 1;38(4):335-343. doi: 10.1097/EJA.0000000000001459.

A description of the surge response and aggregated data outcomes in Scandinavian countries was published in https://onlinelibrary.wiley.com/doi/10.1111/aas.13983.

UPDATE 13 Nov 2024:

ADDITIONAL SUMMARY - EXTENDED INCLUSION PERIOD AND ADDITION OF LONG-TERM OUTCOMES, AND CRITICALLY ILL PATIENTS WITH INFLUENZA AND VIRAL PNEUMONITIS Due to the continued influx of patients requiring intensive care due to COVID-19, we extended the inclusion period to 31 Dec 2022. Thus this new cohort will include all patients admitted to ICUs in Sweden from 6 March 2020 to 31 Dec 2022.

We will investigate short (30day mortality) and long-term outcomes (365d mortality and cardiovascular complications) of patients admitted to Swedish ICUs with confirmed SARS-CoV-2 infection and COVID-19 disease.

In international research, the long-term effects of ICU-requiring COVID-19 are now highly topical. Long-term follow-up exceeding one year has not yet been conducted on any Swedish material. To concretely understand the actual implications of long-term outcomes, it is becoming almost standard to compare this patient group to ICU-requiring influenza + viral pneumonitis patients to some extent. We have applied for and obtained ethical approval to include this group as a potential comparator to COVID-19 patients.

However, such comparisons require careful consideration of potential confounders, such as patient characteristics and socioeconomic factors.

It is therefore crucial to both establish the disease burden for the population and relate it to a comparable patient group. Ethical approval and national data linkage approvals have now been obtained to extract this data from Statistics Sweden and the Swedish National Board of Health and Welfare registries. Data linkage was completed in October 2024.

DETAILED DESCRIPTION:
Previous studies reporting outcomes for COVID-19 patients admitted to intensive care units (ICUs) have been hampered by right-censoring after short observation periods. None have reported 30-day mortality rates and the vast majority of studies have substantial proportions of undischarged patients at the time of follow-up. The lack of follow-up at least to ICU discharge may cause bias in reported mortality rates. Further, national data on critically ill patients have not been previously published.

UPDATE 26 Feb 2022: A number of large, cohort studies including national population outcomes have now been published.

This is a registry-based cohort study of all adult patients (≥18 years) admitted to Swedish Intensive Care Units with confirmed SARS-CoV-2 infection and COVID-19 disease during the first 2 months of the 2020 pandemic. The Swedish Intensive Care Registry (SIR) collects data on patients admitted to all Swedish ICUs, with 100% coverage since 2019. Thus, SIR is able to report on outcomes in a national intensive care population without selection. Little is known about the epidemiology of COVID-19 infections in Sweden, which has one of the world's highest life expectancies and a significant burden of comorbidity. Coupled with Sweden's 'relaxed' approach to COVID-19 pandemic management, health care outcomes are understandably under question.

The main goal is to describe demographic characteristics, coexisting conditions, treatments and outcomes among critically ill patients with COVID-19. A secondary goal is to identify independent risk factors associated with increased mortality for these patients.

ADDITIONAL SUMMARY updated 20 October 2021 Due to the continued influx of COVID-19 patients in ICUs in Sweden throughout 2020 and 2021, we extended of our sample size to encompass all patients admitted up to 30 June 2021 (previously 6 May 2020).

We aim to investigate short- and long-term outcomes including mortality and the incidence of new cardiovascular and respiratory diagnoses up to one year after inclusion.

On 22 mar 2021 we received ethical committee approval for these extensions.

UPDATE 31 October 2024 We have sought and obtained ethical approval to extend the inclusion period to 31 Dec 2022. Data linkage with the Swedish causes of death registry, Swedish Death Registry, Swedish National Patient Registry was approved and data obtained on 11 Oct 2024. This data will be used to investigate long-term outcomes including mortality, new cardiovascular and respiratory diagnoses. Compared to the update on 20 Oct 2021, we will investigate outcomes at longest follow-up, rather than at one year.

We have also sought and obtained ethical approval to expand the cohort to include all patients with viral pneumonitis admitted to Swedish ICUs between 1 jan 2005-31 dec 2022. This cohort will act as a comparator group to COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* COVID-19 disease

Exclusion Criteria:

* No Swedish personal identity number
* 'Opt out' from Swedish Intensive Care Registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years)
  admitted to Swedish Intensive Care Units with confirmed SARS-CoV-2 infection and COVID-19 disease during the first 2 months of the 2020 pandemic (6 March-6May2020).
Sampling Method: Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  all-cause
365-day mortality | 365 days (additional outcome added Oct 2021 after additional approval from ethical committee)
  all-cause

SECONDARY OUTCOMES:
ICU mortality | 30 days
  all cause
Morbidity | up to 365 days after study inclusion
  Cardiovascular and Respiratory Diseases

OTHER OUTCOMES:
Mortality at longest follow-up | 6 Mar 2020 to 31 Dec 2022
  All cause mortality at longest follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesia and Intensive Care, Linkoeping University Hospital, Region Östergötland, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Unidentified data will be shared conditional upon application to the CI

REFERENCES:
- [Derived] Chew MS, Blixt PJ, Ahman R, Engerstrom L, Andersson H, Berggren RK, Tegnell A, McIntyre S. National outcomes and characteristics of patients admitted to Swedish intensive care units for COVID-19: A registry-based cohort study. Eur J Anaesthesiol. 2021 Apr 1;38(4):335-343. doi: 10.1097/EJA.0000000000001459. PMID 33534266